## September 24, 2020

I do not have the study protocol or informed consent. The study was terminated due to insufficient enrollment. No study data are available. All study protocols and informed consent have been deleted and cannot be retrieved at this time.

Rachael Overcash, MD, MPH

MedStar Research Institute

Washington, DC